CLINICAL TRIAL: NCT03574974
Title: Neurofeedback of Amygdala Activity for Post-traumatic Stress Disorder (PTSD)
Brief Title: Neurofeedback of Amygdala Activity for Post-traumatic Stress Disorder
Acronym: PTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended prematurely
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000022668; 1R61MH115110-01A1 (NIH)
Record Dates: First submitted 2018-06-07; First posted 2018-07-02 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Neurofeedback
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will receive either an experimental feedback intervention or a control feedback intervention. Participants who receive the control feedback intervention will be offered to return to receive the experimental feedback intervention upon completion of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be blind to group assignment (experimental feedback intervention or control feedback intervention). The outcome assessor will be blind to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Feedback Intervention (Experimental): Participants receive real-time feedback during fMRI scans that the investigators believe may help them learn to control their PTSD symptoms.
  Interventions: Device: Experimental Feedback
- Control Feedback Intervention (Placebo Comparator): Participants receive real-time feedback during fMRI scans that the investigators do not believe can help their PTSD symptoms.
  Interventions: Device: Control Feedback

INTERVENTIONS:
Device: Experimental Feedback — Feedback is presented in the form of a line graph that is updated every 2 seconds throughout the scan to indicate activity in the target area. A red diamond will indicate periods of symptom provocation, during which participants are exposed to symptom-provoking auditory stimuli in the form of personalized trauma scripts and sound clips. A blue arrow will indicate periods of down-regulation, where participants will try to bring the feedback line down as much as possible (by trying to decrease their fear/anxiety). The investigators believe that this feedback may help participants learn to control their PTSD symptoms.
  Participants will attend a total of 18 feedback scans over the course of 3 sessions.
  Arms: Experimental Feedback Intervention
Device: Control Feedback — Feedback is presented in the form of a line graph that is updated every 2 seconds throughout the scan to indicate activity in the target area. A red diamond will indicate periods of symptom provocation, during which participants are exposed to symptom-provoking auditory stimuli in the form of personalized trauma scripts and sound clips. A blue arrow will indicate periods of down-regulation, where participants will try to bring the feedback line down as much as possible (by trying to decrease their fear/anxiety). The investigators do not believe this feedback can help participants' PTSD symptoms.
  Participants will attend a total of 18 feedback scans over the course of 3 sessions.
  Arms: Control Feedback Intervention

SUMMARY:
The primary purpose of this study is to investigate the efficacy of neurofeedback (NF) of real-time functional magnetic resonance imaging (rt-fMRI) data of the amygdala with regards to the reduction of post-traumatic stress disorder (PTSD) symptoms.

A secondary purpose of this study is to use fMRI as a method of investigating brain function in individuals with PTSD. This study approach provides a tool for probing the neurobiology of PTSD by (1) testing the critical role of the amygdala in this disorder, and by (2) examining how amygdala connectivity is related to both amygdala regulation and clinical symptoms.

DETAILED DESCRIPTION:
In pursuit of the overarching goals of this study, the investigators aim to:

* determine if an experimental feedback intervention increases control over the region of interest (the amygdala) more than a control feedback intervention in which participants receive feedback that is unassociated with their PTSD symptoms.
* determine if an experimental feedback intervention results in clinical improvements in PTSD symptoms relative to a control feedback intervention, and examine whether these improvements correlate with improved control over the amygdala.
* determine if an experimental feedback intervention results in changes in resting state connectivity to the amygdala, and whether these changes correlate with symptom improvement and an improved ability to regulate the amygdala.

ELIGIBILITY:
Inclusion Criteria

* Ages 18 and up
* Diagnosis of chronic PTSD, as established by the Clinician Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V; CAPS-5)
* Ability to give signed, informed consent in English
* Normal or corrected-to-normal vision
* Participants who are on a stable dose of selective serotonin reuptake inhibitor (SSRI) antidepressants for 2 months (3 months if they are on sertraline), or who have been un-medicated for at least 2 months, will be allowed to participate in this study
* At the time of recruitment, patients must have no intention of changing their medication or psychotherapy during the 2.5-month period of the intervention
* Research group must be able to identify a trauma-related target region in or immediately adjacent to the amygdala

Exclusion Criteria

* Any primary psychiatric diagnosis of a current major mood disorder, psychotic disorder, autism, mental retardation, or DSM-5 substance use disorder of mild or greater severity (2 or more symptoms) in the past 30 days. Comorbid mood and anxiety disorders will be permitted if they are not the primary focus of clinical attention
* Any history of psychosis or mania
* Active suicidality within past year, or history of suicide attempt in past 2 years
* Any contraindication to MRI scanning (severe claustrophobia, ferromagnetic metal in body, etc.)
* Pregnancy
* Any unstable medical or neurological condition
* Any history of severe past drug dependence (i.e., a focus of clinical attention or a cause of substantial social or occupational difficulty)
* Any history of brain surgery, of penetrating, neurovascular, infectious, or other major brain injury, of epilepsy, or of other major neurological abnormality (including a history of traumatic brain injury [TBI] with loss of consciousness for more than 24 hours or posttraumatic amnesia for more than 7 days)
* Significant hearing loss or severe sensory impairment
* Any psychotropic medication other than a stable dose of selective serotonin reuptake inhibitors (SSRIs)
* Any change in accepted psychotropic medication within the past 2 months
* Active engagement in cognitive-behavioral therapy or any evidence-based PTSD psychotherapy (Cognitive Processing Therapy [CPT], Prolonged Exposure [PE], Eye Movement Desensitization and Reprocessing [EMDR]) initiated within the past 3 months; continuation of established maintenance supportive therapy will be permitted
* Enrollment in another research study testing an experimental/clinical/behavioral intervention intended to affect symptoms initiated within the last 2 months, or intended enrollment within the next 2.5 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Harpaz-Rotem, PhD, Principal Investigator — Yale University School of Medicine, VA; Michelle Hampson, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale School of Medicine, New Haven, Connecticut
  - VA Connecticut Healthcare System - West Haven Campus, West Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Feedback Intervention: Participants receive real-time feedback during fMRI scans that the investigators believe may help them learn to control their PTSD symptoms.
  Experimental Feedback: Feedback is presented in the form of a line graph that is updated every 2 seconds throughout the scan to indicate activity in the target area. A red diamond will indicate periods of symptom provocation, during which participants are exposed to symptom-provoking auditory stimuli in the form of personalized trauma scripts and sound clips. A blue arrow will indicate periods of down-regulation, where participants will try to bring the feedback line down as much as possible (by trying to decrease their fear/anxiety). The investigators believe that this feedback may help participants learn to control their PTSD symptoms.
  Participants will attend a total of 18 feedback scans over the course of 3 sessions.
- Control Feedback Intervention: Participants receive real-time feedback during fMRI scans that the investigators do not believe can help their PTSD symptoms.
  Control Feedback: Feedback is presented in the form of a line graph that is updated every 2 seconds throughout the scan to indicate activity in the target area. A red diamond will indicate periods of symptom provocation, during which participants are exposed to symptom-provoking auditory stimuli in the form of personalized trauma scripts and sound clips. A blue arrow will indicate periods of down-regulation, where participants will try to bring the feedback line down as much as possible (by trying to decrease their fear/anxiety). The investigators do not believe this feedback can help participants' PTSD symptoms.
  Participants will attend a total of 18 feedback scans over the course of 3 sessions.
Period: Overall Study
Arm/Group | Experimental Feedback Intervention | Control Feedback Intervention
Started | 15 | 12
Completed | 14 | 11
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Feedback Intervention | Control Feedback Intervention | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Customized [Mean (Standard Deviation); unit: years] | 40.2 (14.27) | 50.36 (12.78) | 44.67 (14.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 11 | 25
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 25
Medication Status [Count of Participants; unit: Participants]
  No psychiatric medication | 4 | 4 | 8
  Antidepressants | 7 | 2 | 9
  Anticonvulsant | 0 | 2 | 2
  Stimulants | 1 | 0 | 1
  Medical Marijuana/Cannabinoids (CBD Oil) | 1 | 3 | 4
  Unknown | 1 | 0 | 1
Clinician-Administered PTSD scale for Diagnostic and Statistical Manual of Mental Disorders, (CAPS-5 [Mean (Standard Deviation); unit: score] — Clinician-Administered PTSD scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) [CAPS-5]). The CAPS5 ranges from 0 (no symptoms) to 80 (maximum score). A higher score is associated with higher severity of PTSD. The score is interpreted as follows: 0-10 = asymptomatic/few symptoms, 11-22 = mild PTSD/sub-threshold PTSD, 23-34 = moderate PTSD/threshold, 35-46 = severe PTSD, and score 47 and above = extreme PTSD.
  score | 33.71 (7.99) | 39.73 (9.27) | 36.36 (8.93)
PTSD Checklist for DSM-5 (PCL-5) [Mean (Standard Deviation); unit: score] — The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Scores 31 and above are indicative of PTSD.
  score | 43.43 (13.42) | 47.45 (14.03) | 45.20 (13.555)
Additional Diagnoses [Count of Participants; unit: Participants]
  Major Depressive Disorder(MDD) | 5 | 5 | 10
  MDD in partial remission | 2 | 2 | 4
  MDD in full remission | 5 | 2 | 7
  Dysthymic Disorder | 0 | 0 | 0
  Obsessive-Compulsive Disorder | 3 | 0 | 3
  Social Phobia | 5 | 3 | 8
  Generalized Anxiety Disorder | 2 | 2 | 4
  Body Dysmorphic Disorder | 2 | 2 | 4
  Panic Disorder with Agoraphobia | 1 | 1 | 2
  Panic Disorder without Agoraphobia | 1 | 3 | 4
  Agoraphobia without History of Panic Disorder | 1 | 0 | 1
  Phobia of Heights | 0 | 1 | 1
  Stratification: high re-experiencing (vs low) | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Control Over the Amygdala
Description: Control over the amygdala will be defined as the change in the blood-oxygen-level dependent (BOLD) signal in the target area (an individually-localized region of interest (ROI) in the amygdala) during down-regulation blocks following symptom provocation relative to rest. Investigators will assess the magnitude of change in control over the amygdala to trauma reminders from baseline to 30-day post treatment follow-up. This measure is based on beta values, which are unitless
Time Frame: baseline; 30 day-day follow up
Measure: Mean (Standard Error); unit: unitless
Arm/Group | Experimental Feedback Intervention | Control Feedback Intervention
Number analyzed (Participants) | 14 | 11
unitless | -0.279 (0.146) | 0.202 (0.167)
Statistical Analysis 1: Comparison: Experimental Feedback Intervention vs Control Feedback Intervention; Test type: Superiority; p = 0.047, t-test, 2 sided

2. Secondary Outcome: Improvements in PTSD Symptoms
Description: Clinical improvement will be defined as the change from baseline at the post-intervention assessments (based on the past-month Clinician-Administered PTSD scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V ) [CAPS-5]). Score ranges from 0 - no PTSD symptoms to a maximum of 80. Higher score is associated with increase severity of PTSD. A change in CAPS score of more than 5 points over the course of treatment is considered a meaningful change and a change of 10 point or more is considered to be a clinically meaningful change.
Time Frame: Baseline; 30-day follow-up
Measure: Mean (Standard Deviation); unit: Average CAPS change score
Arm/Group | Experimental Feedback Intervention | Control Feedback Intervention
Number analyzed (Participants) | 14 | 11
Average CAPS change score | 8.786 (9.744) | 10.545 (13.441)

3. Secondary Outcome: Improvements in PTSD Symptoms
Description: as for outcome 2
Time Frame: Baseline; 60-day follow-up
Measure: Mean (Standard Deviation); unit: Average change in CAPS scores
Arm/Group | Experimental Feedback Intervention | Control Feedback Intervention
Number analyzed (Participants) | 14 | 11
Average change in CAPS scores | 13.286 (9.934) | 9.364 (13.246)

4. Secondary Outcome: Number of Participants With Changes in Resting State Connectivity to the Amygdala
Description: The number of participants with a significant whole brain change in seed region connectivity to the amygdala from pre- to post-intervention will be assessed in the blood-oxygen-level dependent (BOLD) signal collected during resting state runs.
Time Frame: Baseline; 60 days follow up.
Population: Due to the COVID-19 suspension of human subject research, resting state date for 60-day post treatment were not available for 4 participants in the experiential group and 1 subject in the control group.
Measure: Number; unit: number of participants with change
Arm/Group | Experimental Feedback Intervention | Control Feedback Intervention
Number analyzed (Participants) | 10 | 10
number of participants with change | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 60 days
Arm/Group | Experimental Feedback Intervention | Control Feedback Intervention
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 0/15 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT03574974/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT03574974/ICF_001.pdf